CLINICAL TRIAL: NCT04266626
Title: Clinical and Psychological Outcomes of Kinesiotaping and Manipulation Therapies in Drooling Management Among Children With Oral Dysphagia
Brief Title: Effectiveness of Kinesiotaping and Manipulation Therapies in Drooling Management Among Children With Oral Dysphagia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isra University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1602-PhD-004
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Drooling
Keywords: dysphagia, drooling, kinsesiotaping therapy, manipulation therapy
MeSH Terms: conditions — Sialorrhea; Deglutition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A kinesiotaping therapy (Experimental): Protocols mentioned in kinesiological taping i.e. 45 minutes will be pursued as with longer sessions children may tire out easily. Taping Technique for lip muscles would be used by cutting 2 "I" tapes according to the structure of lip muscles.The tape will be fixed in the center of the mouth on the upper lip, will be placed on an open mouth and a 10% tension will be given to the paper. The tape will then end at the corner of the upper lip. Kinesiotape wouldn't be placed on the lips. The second tape piece will be fixed to the center of the lower lip.The edges of the tape should overlap slightly.
  The other piece of tape will be placed under chin (base of tongue) on sub mandibular triangle, inside the jaw line on the base of the tongue. A strip 1-1 ½ inch long will be cut, and then will further be cut in half such that the stretch is horizontal. It will be anchored in the middle on sub mandibular triangle. Paper off the tension to both sides.
  Interventions: Other: kinesiotaping therapy
- Group B Oral Motor Manipulation therapy (Active Comparator): For the oral motor manipulation technique CP chair will be required to maintain the good sitting posture of children. Trunk will be in upright position with cut out lap board of the CP chair. Hips, knees and ankles would be flexed to 90 degrees. Shoulders and arms will be rested in symmetrical manner by keeping them rested in lap board and foot rest will be used to rest the feet tightly to control movement and maintain good posture. Each child would be taken for 12 weeks of therapy with three sessions per day of 15 minutes each. Oral motor manipulation like tapping protocols would be used for 45 minutes; slow, even rhythmic pressure will be applied around lip muscle and base of tongue muscle, keeping in view the comfort level of patient.
  Training to do manipulation exercises will be given to the parents of children with CP at .
  Interventions: Other: oral motor manipulation therapy

INTERVENTIONS:
Other: kinesiotaping therapy — Kinesiotaping is a new therapeutic technique that gives support to the lip and tongue base muscles without restricting range of motion or blood flow.
  Arms: Group A kinesiotaping therapy
Other: oral motor manipulation therapy — Manipulation therapy include tapping and massage of oral motor muscles including orbicularis oris and base of tongue.
  Arms: Group B Oral Motor Manipulation therapy

SUMMARY:
Children suffering from neurological problems may have a common problem of drooling and dysphagia.There is high prevelance of neurological disorders in developing countries including Pakistan.Parents of children with disability are highly stressed and burdenised while taking care of their children.there is a need to overcome the drooling and dysphagia problems with effective interventions.

DETAILED DESCRIPTION:
There is no clear consensus that which interventions are safe and effective and hard to decide about the effective intervention for drooling management. This will help the parents, therapist and children to manage their feeding problems effectively, hence improve quality of life of parents and children.There is also scarcity of well designed randomized controlled trails and limited published literature on the usefulness of the kinesiotape for management of drooling in children with oral dysphagia, this study will be conducted in an attempt to evaluate the same. There is also a lack of comparative studies to evaluate the effectiveness of traditional oral motor therapies and kinesiotaping therapy.

speech pathologists and help them in managing drooling effectively by using the best effective therapeutic approach. This study will also add up evidence-based knowledge to existing literature

ELIGIBILITY:
Inclusion Criteria:

* • Both male and female children with different non degenerative neurological disabilities ( cerebral palsy, traumatice brain injury, childhood stroke) and having oral phase dysphagia.

  * Age between 3-15 years.
  * Those who will have drooling severity rating of ≥ 4 on modified Teacher's drooling scale.
  * Child who can comprehend simple verbal commands and on 3 words sentence level speech
  * Have good head control.
  * Parents and care givers of children with drooling and oral phase dysphagia will also be included in the study

Exclusion Criteria:

* Those children who would have structural abnormality of respiratory system.
* Corrected or uncorrected cleft palate or cleft lip.
* Wounds around the lips.
* Recent surgery, and medication or on any treatment to control drooling would be excluded from the study.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
severity and frequency of drooling will be measured at baseline and at the end of 24 weeks of therapy | 24 weeks
  half of both groups will be intervene for 12 weeks first and other half groups after 12 weeks, so total 24 weeks will be required for whole group to be intervene

CONTACTS AND LOCATIONS:
Overall Officials: Romana Pervez, PhD, Principal Investigator — helping hand Institute of Rehabilitation Sciences Mansehra
Locations (1):
- Romana Pervez, Abbottabad, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No